CLINICAL TRIAL: NCT00346853
Title: Clinical Interventions Against Stargardt Macular Dystrophy: Phase 1 Pilot Study of 4-MP as an Inhibitor of Dark Adaptation
Brief Title: Phase 1 Pilot Study of 4-MP to Treat Stargardt Macular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Dr. Randall Olson, Chair, Department of Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-MP Dark Adaptation Inhib.
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Macular Dystrophy, Corneal
Keywords: Dark adaptation inhibition; Stargardt macular dystrophy; 4-Methylpyrazole (4-MP); Antizol; Fomepizole
MeSH Terms: conditions — Corneal Dystrophies, Hereditary; Stargardt Disease | interventions — Fomepizole; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: 4-Methylpyrazole
- 2 (Placebo Comparator): saline
  Interventions: Other: saline

INTERVENTIONS:
Drug: 4-Methylpyrazole — 15 mg/kg dose
  Arms: 1
Other: saline
  Arms: 2

SUMMARY:
The purpose of this study is to investigate whether taking 4-methylpyrazole (4-MP, fomepizole, Antizol™) inhibits dark adaptation of the eye. In other words, we are testing if 4-MP slows the processing of vitamin A derivatives in the eye. By slowing down these processes, individuals with Stargardt disease may have better chances of saving their remaining vision. 4-MP has been shown to slow dark adaptation in animals, and is FDA approved for human use to treat individuals with methanol or ethylene glycol (antifreeze) poisoning by shutting down the body's ability to process alcohols. This medication has an excellent safety profile and has been reported to have no short-term or long-term side effects, as long as patients refrain from any alcohol while the medication is in the body. A single dose of 4-MP remains in the body for about 12 hours, and therefore, it may inhibit dark adaptation of your eyes for up to 12 hours. Studying the effects of 4-MP may lead to effective medical treatment to save Stargardt patients' vision, and may also have similar effects in other macular degenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* All nonpregnant, nonlactating adults with normal vision in both eyes

Exclusion Criteria:

* Previous ocular pathologies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-11; Primary Completion 2006-05 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Dark adaptation inhibition measured 30 minutes after drug infusion using Goldman-Weeker adaptometer. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Bernstein, M.D., Ph.D., Principal Investigator — University of Utah
Locations (1):
- Moran Eye Center, University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Jurgensmeier C, Bhosale P, Bernstein PS. Evaluation of 4-methylpyrazole as a potential therapeutic dark adaptation inhibitor. Curr Eye Res. 2007 Oct;32(10):911-5. doi: 10.1080/02713680701616156. PMID 17963111